CLINICAL TRIAL: NCT05022719
Title: A Prospective Single-center Pilot Study Evaluating the Technical Feasibility of Mucosal Staining During Colon Capsule Endoscopy (CCE) Procedure in Colorectal Cancer (CRC) High Risk Population, When Using MB-MMX (SPICE Study)
Brief Title: Technical Feasibility Evaluation of Mucosal Staining During Colon Capsule Endoscopy (CCE) Procedure in Colorectal Cancer (CRC) High Risk Population, When Using MB-MMX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT20062
Record Dates: First submitted 2021-08-12; First posted 2021-08-26 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Polyp, Colonic
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, non-randomized clinical trial designed to evaluate the technical feasibility during CCE procedure, when using MB-MMX as a contrast- enhancement technique of mucosal staining in CRC high risk population.
  Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg). An experienced Gastroenterologist will read the CCE procedure and complete a subjective questionnaire, to evaluate mucosal enhancement during a CCE procedure, when using MB-MMX as a contrast-enhancement technique.
  The technical feasibility will be evaluated by:
  1. The percent of colonic polyps which have a visible contrast to the healthy colonic mucosa during CCE.
  2. The interference level of detrimental effects on the visualization of the colonic mucosa during CCE, due to use of MB-MMX per colonic segment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PillCam Colon2 procedure with MB-MMX (Experimental): PillCam Colon2 procedure with MB-MMX
  Interventions: Device: PillCam Colon2 procedure with MB-MMX

INTERVENTIONS:
Device: PillCam Colon2 procedure with MB-MMX — Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg). An experienced Gastroenterologist will read the CCE procedure and complete a subjective questionnaire, to evaluate mucosal enhancement during a CCE procedure, when using MB-MMX as a contrast-enhancement technique.

SUMMARY:
A prospective, single-center, single-arm, non-randomized, post-market pilot study evaluating the technical feasibility of mucosal staining during COLON2 Capsule Endoscopy (CCE) procedure in population at high risk for Colorectal Cancer (CRC), when using MB-MMX (Methylene Blue).

Up to 15 subjects will be enrolled in 1 center located in Spain. Study duration- up to 10 months from study approval.

DETAILED DESCRIPTION:
Single-center, prospective, non-randomized clinical trial designed to evaluate the technical feasibility during CCE procedure, when using MB-MMX as a contrast- enhancement technique of mucosal staining in CRC high risk population.

Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg). An experienced Gastroenterologist will read the CCE procedure and complete a subjective questionnaire, to evaluate mucosal enhancement during a CCE procedure, when using MB-MMX as a contrast-enhancement technique.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ages 45-75 years
2. Subject is classified as being at high risk for CRC due to one (or more) of the following risk factors:

   * A personal history of colorectal polyps
   * A first-degree family history of colorectal cancer
   * Family/personal inherited syndrome (Lynch syndrome, Familial adenomatous polyposis {FAP}, other inherited syndromes linked to colorectal cancer)
   * Subject with currently suspected or diagnosed rectal bleeding, including positive FIT or positive fecal DNA test
   * Subjects under surveillance for CRC (last OC≥1.5 years)
3. Subject is willing and able to participate in study procedures, understand and sign the informed consent

Exclusion Criteria:

1. Subject has a previous history or suspicion of inflammatory bowel or Crohn's disease, ulcerative Colitis or indeterminant Colitis
2. Subject has congestive heart failure or recent myocardial infarction (<3month)
3. Subject with moderate/severe renal disease and/ or severe hepatic impairment
4. Subject has uncontrolled diabetes
5. Subject has a severe, life-threatening disease
6. Subject with known gastrointestinal motility disorders
7. Subject has known delayed gastric emptying
8. Subject has undergone surgery of the luminal gastrointestinal (GI) tract, from esophagus to the rectum, other than uncomplicated appendectomy or cholecystectomy.
9. Subject with any current condition believed to have an increased risk of capsule retention such as suspected or known bowel obstruction or pseudo-obstruction, stricture, or fistula (symptoms such as severe abdominal pain with accompanying nausea or vomiting)
10. Subject with dysphagia, any swallowing disorder, or any major gastrointestinal motility disorder
11. Subject has a history of inadequate bowel preparation for colon imaging with colonoscopy, CTC, CCE, or DCBE (self-reporting)
12. Subject with known or suspected constipation history as defined by the following: as needing the use of medication (prescription or OTC) for management of constipation, or fewer than 3 BM/week regardless of medication use
13. Subject with a cardiac pacemaker or other implanted electromedical device
14. Subject with planned MRI examination within 7 days after ingestion of the capsule
15. The subject is taking antidepressant medicine or a medicine for psychiatric illness, such as:

    * selective serotonin reuptake inhibitor (SSRI)- as fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, escitalopram and zimeldine; bupropion, venlafaxine, mirtazapine, clomipramine, buspirone
    * medicines classified as Monamine Oxidase Inhibitors (often used for treating depression).
16. Subject has glucose-6-phosphate dehydrogenase (G6PD) deficiency and/or allergic to peanut/soya
17. Subject consumes any of the medicinal products which interacts with MB-MMX, as per MB-MMX label and Investigator's discretion.
18. Subject with allergies or known contraindication to the device, medications or preparation agents used in the procedure as described in the relevant instructions for use/package inserts.
19. Subject use of opioid medication on a regular basis and requires medication to treat opioid induced constipation
20. Subject currently participating in another gastrointestinal clinical study (investigational drug or device) that might interfere with results of study
21. Females who are pregnant or breastfeeding at time of bowel prep
22. Any condition which precludes compliance with study and/or device instructions based on the clinical judgment of the investigator
23. Subject who is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity)
24. Medtronic employees

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Split Dose: Subjects will undergo a bowel preparation (split dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg).
- PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Single Dose: Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg).
Period: Overall Study
Arm/Group | PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Split Dose | PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Single Dose
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PillCam Colon2 With Methylene Blue (MB-MMX) Split Dose: Subjects will undergo a bowel preparation (split dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg) as bowel preparation for PillCam Colon2 Capsule Endoscopy (CCE)
- PillCam Colon2 With Methylene Blue Single Dose: Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg) as bowel preparation for PillCam Colon2 Capsule Endoscopy (CCE)
- Total: Total of all reporting groups
Arm/Group | PillCam Colon2 With Methylene Blue (MB-MMX) Split Dose | PillCam Colon2 With Methylene Blue Single Dose | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [57 to 74] | 58.3 [49 to 68] | 62.9 [49 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 5 | 3 | 8
BMI [Mean (Full Range); unit: kg/m^2] — kg/m^2
  kg/m^2 | 27.3 [26.1 to 34] | 26.6 [22.7 to 29.1] | 27.1 [22.7 to 34]

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Colonic Polyps Which Have a Visible Contrast to the Healthy Colonic Mucosa During Colon Capsule Endoscopy (CCE)
Description: The percent of colonic polyps which have a visible contrast to the healthy colonic mucosa during CCE, as indicated by an experienced reader, using the subjective reader questionnaire (For each polyp - was there a contrast between the polyp and the healthy mucosa? Yes/No), out of the examined polyps
Time Frame: During the CCE procedure
Population: All subjects were included in the Per Protocol Analysis (N=8); 30 total polyps were visualized across the 8 patients.
Measure: Number (95% Confidence Interval); unit: percentage of polyps with contrast
Units Other Than Participants: # of Polyps
Groups:
- PillCam Colon2 Procedure With MB-MMX Split Dose: PillCam Colon2 procedure with MB-MMX: Subjects will undergo a bowel preparation (split dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg). An experienced Gastroenterologist will read the CCE procedure and complete a subjective questionnaire, to evaluate mucosal enhancement during a CCE procedure, when using MB-MMX as a contrast-enhancement technique.
- PillCam Colon2 Procedure With MB-MMX Single Dose: PillCam Colon2 procedure with MB-MMX: Subjects will undergo a bowel preparation (single dose, 4L PEG), including 200 mg Methylthioninium chloride, corresponding to eight 25 mg MB-MMX tablets and 1 tab of Resolor (Prucalopride 1mg). An experienced Gastroenterologist will read the CCE procedure and complete a subjective questionnaire, to evaluate mucosal enhancement during a CCE procedure, when using MB-MMX as a contrast-enhancement technique.
Arm/Group | PillCam Colon2 Procedure With MB-MMX Split Dose | PillCam Colon2 Procedure With MB-MMX Single Dose
Number analyzed (Participants) | 5 | 3
Number analyzed (# of Polyps) | 24 | 6
percentage of polyps with contrast
  Overall % Polyps with Contrast | 58.3 [36.6 to 77.9] | 66.7 [22.3 to 95.7]
  % Cecum Polyps | 0 [0 to 0] | 0 [0 to 0]
  % Ascending Polyps | 100 [29.2 to 100] | 0 [0 to 0]
  % Transverse Polyps | 50 [1.3 to 98.7] | 100 [100 to 100]
  % Descending Polyps | 66.7 [9.4 to 99.2] | 100 [100 to 100]
  % Rectal Polyps | 50 [24.7 to 75.4] | 66.7 [9.4 to 99.2]

2. Primary Outcome: The Interference Level of Detrimental Effects on the Visualization of the Colonic Mucosa During Colon Capsule Endoscopy (CCE), Due to Use of MB-MMX Per Colonic Segment.
Description: The interference level of detrimental effects on the visualization of the colonic mucosa during CCE, due to use of MB-MMX per colonic segment. Detrimental effect will be considered as any observation, such as an excessive blue dye deposit, dark and dim appearance of the tissue, interfering with tissue visualization and will be evaluated on a scale from 1 (no interference) to 5 (high interference) to evaluate the level of interference, using a subjective reader questionnaire.
Time Frame: During CCE
Population: All subjects were included in the per protocol analysis set.
Measure: Mean (Standard Deviation); unit: score on a scale of 1 to 5
Arm/Group | PillCam Colon2 Procedure With MB-MMX Split Dose | PillCam Colon2 Procedure With MB-MMX Single Dose
Number analyzed (Participants) | 5 | 3
score on a scale of 1 to 5
  All Segments | 1.2 (0.4) | 4.8 (1)
  Cecum | 1.2 (0.4) | 3.3 (1.2)
  Ascending | 1.2 (0.4) | 1.7 (0.6)
  Transverse | 1.2 (0.4) | 1.3 (0.6)
  Descending | 1.3 (0.5) | 1 (0)
  Rectum | 1 (0) | 1.7 (0.6)

3. Primary Outcome: Subjects With Polyps Visualized During Colon Capsule Endoscopy (CCE)
Description: Count of Subjects with Polyps visualized during Colon Capsule Endoscopy (CCE)
Time Frame: During CCE
Population: All subjects were included in the Per Protocol Analysis (N=8)
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Split Dose | PillCam Colon2 Procedure With Methylene Blue (MB-MMX) - PEG Single Dose
Number analyzed (Participants) | 5 | 3
Participants | 4 | 2

4. Secondary Outcome: To Evaluate the Safety of CCE Procedure While Using MB-MMX.
Description: All AEs will be reported by number, type, relatedness (device/procedure), seriousness, severity and duration. All AEs will be captured, regardless of severity.
Time Frame: Evaluated for each patient enrolled from day -1 prior to the procedure (start of bowel prep intake) until day 5-9 after the procedure (end of follow-up).
Population: All enrolled subjects were included in the safety analysis.
Measure: Number; unit: Events
Arm/Group | PillCam Colon2 Procedure With MB-MMX Split Dose | PillCam Colon2 Procedure With MB-MMX Single Dose
Number analyzed (Participants) | 5 | 3
Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected for all enrolled subjects at the start of the bowel preparation, at day (-1), until the follow-up phone call (visit 3). Medical care will be provided, as defined in the informed consent, for any AE related to study participation, if needed.
Description: Per ISO14155:2020: Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated
Arm/Group | PillCam Colon2 Procedure With MB-MMX Split Dose | PillCam Colon2 Procedure With MB-MMX Single Dose
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT05022719/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT05022719/SAP_001.pdf